CLINICAL TRIAL: NCT07007923
Title: Recruitment of the Diaphragm and Sternocleidomastoid Muscle During Loaded Inspiration on Varying Sitting Support in Healthy Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, LIU FANG, PHD student, Hong Kong Metropolitan University
Other Study IDs: No.HE-OT2023/13
Record Dates: First submitted 2025-05-10; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Diaphragm
Keywords: Diaphragmatic thickening fraction; Sternocleidomastoid muscles; inspiratory pressure

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a cross-sectional obsessional study.

This study explores how different sitting conditions affect two important muscles-the diaphragm and the sternocleidomastoid (SCM)-work during breathing exercises. The diaphragm is the main muscle for breathing, while the SCM helps when taking deeper breaths. Understanding how these muscles interact while sitting under various conditions can help improve breathing training techniques.

The study's objectives are (1) to investigate the relationship between diaphragm thickness fraction with 4 different sitting conditions during loaded inspiration among healthy adults and (2) To investigate the relationship between SCM activity with 4 different sitting conditions during loaded inspiration among healthy adults.

This research will conduct healthy adults, who will be instructed to breathe against resistance provided by the IMT while sitting on four different conditions: a regular chair, a soft pad with feet on the ground, a soft pad with feet on two additional soft pads, and a single soft pad with both feet on one pad. By using ultrasound to measure how thick the diaphragm gets and surface electromyography (sEMG) to track SCM activity, the data will be gathered on how these muscles function under different conditions.

The goal is to find out if sitting on unstable surfaces, like soft pads, can enhance diaphragm use compared to a stable chair. These surfaces may change how effectively the diaphragm and SCM work together. This research could lead to better recommendations for inspiratory muscle training (IMT), which helps strengthen these muscles, especially for people with breathing difficulties.

By identifying how posture influences muscle recruitment during breathing exercises, hoping to contribute valuable insights that can improve rehabilitation programs for individuals with respiratory conditions.

DETAILED DESCRIPTION:
Participant information sheets and consent form will be given and explained to participants prior to experiment. To ensure measurement consistency, one standardized assessor will be employed. Demographic data, including age, sex, exercise habit, and smoking history will be recorded. Health-related quality of life will be quantified by SF-12. Participants who score below 50 in PCS or MCS will be excluded from our study.

All eligible participants will undertake a standard spirometry test to obtain forced vital capacity (FVC), forced expiratory volume in one second (FEV1). Spirometry test will be performed 3 times, in accordance with guidelines recommended by the American Thoracic Society. Participants with findings of obstructive or restrictive disorders will be excluded. MIP will be obtained by a threshold device (S1breathe K5) under standard instruction. Before measuring MIP, specific instructions guiding participants to focus on diaphragm breathing will be instructed (one hand positioned on the subcostal region and allow air to go to the lower part of the chest where your hand is placed) to allow participants aware of the use of diaphragm during trials, therefore they can subconsciously deploy the technique in the subsequent trials. Participants will be allowed to perform 3 times (with nose-clip applied), with the best MIP will be recorded. The thickness of right diaphragm and SCM activity at maximum inspiration, maximum expiration, end-tidal inspiration, end-tidal expiration, and MIP were measured by ultrasonography and sEMG respectively.

Participants will then be instructed to perform IMT in different conditions in a randomized order, completing 4 sets 15 breaths, with a rest period of 5 mins between sets. 50% MIP will be calibrated at the POWERbreathe device with respect to each participant prior IMT. During each inspiratory pressure-targeted breath, simultaneous sEMG recording on the right SCM and ultrasonography of right hemi-diaphragm will be conducted. Participants's subjective exertion level will be recorded by Borg's Rate of Perceived Exertion Scale at the end of each set of recordings.

The POWERbreathe device requires 5 breaths to meet the targeted load. Following the manufacturer's instructions, participants will be instructed to perform with a sharp inspiration lasting 1-2s at each breath for reaching the required load. Each participant will be requested to complete 15 breaths, but only the data from 6th to 15th breaths will be included for analysis. The whole duration will take around 90 minutes. Password code will be used to guarantee anonymity and confidentiality for the data obtained.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-35 years - No recent thoracic surgery in the past 6 months
* Absence in history of chronic respiratory illness
* Able to breathe spontaneously
* Conscious, able to follow instructions on the use of IMT device

Exclusion Criteria:

* with known cardiovascular, pulmonary or musculoskeletal disorders that would limit their functional capacity (E.g. Asthma, COPD)
* presence with respiratory symptoms over past 2 weeks
* pregnancy
* malignancy
* presence of neurological disorders (e.g. ALS, stroke)
* PCS/ MCS in SF-12 scores below 50
* Findings in spirometry suggesting presence of obstructive or restrictive disorders

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: aged 18-35 healthy young adults
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-06-19 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Diaphragmatic thickening fraction | Through study completion, an average of 1 year
  Diaphragmatic thickening fraction is determined by "(thickness of the diaphragm at end inspiratory - thickness at end expiratory)/thickness at end expiratory". Diaphragmatic thickness will be measured by ultrasonography.

SECONDARY OUTCOMES:
Muscle activation of the sternocleidomastoid muscle | Through study completion, an average of 1 year
  Surface electromyography will be used to measure accessory inspiratory muscle (sternocleidomastoid muscles) activity during each inspiratory muscle training intensity.
Borg's scale | Through study completion, an average of 1 year
  The Borg scale is widely used for measuring perceived exertion during physical activity. It can gauge how hard individuals are exerting while taking into account the individual's heart rate, breathing effort, and fatigue level. Participant's subjective experience would also gauge the score of the scale. The Borg RPE scale would be used to measure exertion during exercise as it has a high correlation with physiological measurements. It is quantified from 0 to 10, where 0 represents no symptoms, and 10 represents the maximum symptoms.

OTHER OUTCOMES:
The Short Form (12) Health Survey | Through study completion, an average of 1 year
  The SF-12 is a multidimensional generic measure of health-related quality of life which is based on items taken from the SF-36 health survey. It is composed of standardized questionnaires which cover 12 items selected from the SF-36.It includes 8 domains, physical functioning, role-physical, role-emotional, mental health, bodily pain, general health, vitality, and social functioning. It is scored to produce 2 summary scores, the physical and mental health summaries (PCS and MCS). Scores above 50 predict a better-than-average health-related quality of life. Scores below 50 are considered as below-average health.

CONTACTS AND LOCATIONS:
Overall Officials: William Tsang, Study Director — Hong Kong Metropolitan University
Locations (1):
- Hong Kong Metropolitan University Jockey Club Institute of Healthcare, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2025-05-09): https://cdn.clinicaltrials.gov/large-docs/23/NCT07007923/Prot_SAP_000.pdf
  • Informed Consent Form: Consent form (2025-05-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT07007923/ICF_001.pdf
  • Informed Consent Form: Information sheet (2025-05-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT07007923/ICF_002.pdf